CLINICAL TRIAL: NCT03568903
Title: Functional Performance in Individuals With Parkinson's Disease: Changes Following 2-month Physiotherapy Intervention in Small Groups and Impact of Disease Progression
Brief Title: Changes in Functional Performance in Individuals With Parkinson's Disease Following 2-month Physiotherapy Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tartu (Other)
Collaborators: Tartu University Hospital (Other)
Responsible Party: Principal Investigator, Kadri Medijainen, Junior research fellow/Assistant of physiotherapy, University of Tartu
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: PD_Comprehensive_PT
Record Dates: First submitted 2018-05-15; First posted 2018-06-26 (Actual); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; Gait; Physical therapy; functional performance; group therapy
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Comprehensive physical therapy intervention in small groups (3 members), altogether 16 sessions were performed during a period of 8 weeks (twice a week). Each session lasted 1 hour.
  Interventions: Other: Comprehensive physical therapy
- Control group (No Intervention): Control group members did not receive any specific intervention during study period, but if needed, medical treatment (medication, it's dosage etc) of Parkinson Disease was changed during study period. They were assigned to individual therapy after the study period.

INTERVENTIONS:
Other: Comprehensive physical therapy — Each session included exercises for posture, strength, range of motion, balance. In addition, different transfers and gait training was performed. Each session began with exercises in laying position (15 minutes), thereafter exercises in sitting were performed for 10 minutes. Then different exercises in standing position were performed for 15 minutes, followed by 10 minutes of gait training. 10 minutes of exercises for manual dexterity and upper limb function ended the session.
  Arms: Intervention group

SUMMARY:
Aim of current study was to evaluate the effect of a 2-month comprehensive physiotherapy intervention on different aspects of functional performance. In addition, progression of PD motor symptoms (using standardized clinical tests for the assesment) was of interest

DETAILED DESCRIPTION:
The aim of current study was to enroll 50 patients with Parkinson's disease (PD) and randomly assign them into intervention and control group. Patients were randomly contacted through the epidemiological database of patients with Parkinson' disease of South-Estonia. 44 participants agreed to come to the baseline assessment including:

* Timed-Up-And-Go Test Battery
* Four square step test
* Physical performance test
* Short Physical Performance
* 10-m walk test
* Grooved Purdue Pegboard test
* Assessment of range of motion In addition, current disease status was assessed using Unified Parkinson Disease Rating Scale, Mini Mental Sate Examination. Further, quality of life was assessed using PDQ-39, hand-writing was recorded using white, squared and striped paper and freezing of gait questionaire (FOG-Q) was administered. Within a week from baseline assessment participants randomly assigned to intervention group, started physiotherapy intervention. The intervention was carried out in small groups (3 people in a group) and was carried out as out-patient physiotherapy during 8 week period. During each week 2 sessions with a length of an hour were scheduled. Within a week of the last therapy session, second assessment was conducted (for control group the second assessment was carried out ten weeks post-baseline assessment.

Third assessment was assigned one year after (then the same assessment was performed, in addition body composition was analysed using DXA), forth assessment an other year later.

During forth assessment 15 members starting in the intervention group and 10 starting in the control group participated.

ELIGIBILITY:
Inclusion Criteria:

1. confirmed diagnosis of idiopathic Parkinson Disease
2. age within the age limits
3. no other untreated medical conditions that might affect gait or postural stability
4. able to walk without assistive device
5. score of Mini Mental State Examination above 24
6. no other neurological conditions in medical anamnesis

Exclusion Criteria:

Not meeting the inclusion criteria

Ages: 60 Years to 81 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2013-02-01 (Actual); Primary Completion 2015-05-15 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
Gait speed during transitioning from sitting to walking and its change as a result of physiotherapy and change over time | it was assessed during all the assessments: at baseline, during second assessment ten weeks later, third assessment was carried out one year later, forth assessment was conducted another year later
  Gait speed was calculated based an the performance of Timed up and Go test
Gait speed during transitioning from standing to walking and its change as a result of physiotherapy and change over time | it was assessed during all the assessments: at baseline, during second assessment ten weeks later, third assessment was carried out one year later, forth assessment was conducted another year later
  Gait speed was calculated based an the performance of Short Physical Performance Battery gait test
"Pure" gait speed and its change as a result of physiotherapy and change over time | it was assessed during all the assessments: at baseline, during second assessment ten weeks later, third assessment was carried out one year later, forth assessment was conducted another year later
  Gait speed was calculated based an the performance of 10 m walk test, with excluding the acceleration and deceleration phase (duration of the intermediate 6-meters was measured and based on that gait speed was calculated

SECONDARY OUTCOMES:
body composition (and changes in it in one year period) | was assessed twice (during third and fourth assessment), with a timeperiod of one year in between
  it was assessed with DXA methodology
Timed-up-and-go test: its change as a result of physiotherapy and change over time | it was assessed during all the assessments: at baseline, during second assessment ten weeks later, third assessment was carried out one year later, forth assessment was conducted another year later
  The duration of Timed up and go test, executed with a turn over both shoulders was used
Four square step test: its change as a result of physiotherapy and change over time | it was assessed during all the assessments: at baseline, during second assessment ten weeks later, third assessment was carried out one year later, forth assessment was conducted another year later
  The duration of Four square step test,was used
Tinetti test: its change as a result of physiotherapy and change over time | it was assessed during all the assessments: at baseline, during second assessment ten weeks later, third assessment was carried out one year later, forth assessment was conducted another year later
  The Tinetti test was executed and the score was used
Range of motion: its change as a result of physiotherapy and change over time | it was assessed during three assessments: at baseline, during second assessment ten weeks later, third assessment was carried out one year later
  Range of motion of major joints (shoulder, hip, knee, ankle) were measured goniometrically. Spinal ROM (including neck) was measured with tapemeasure, aswell as the excursion of the ribcage during maximal inspiration and expiration
Assessment of handwriting:its change as a result of physiotherapy and change over time | it was assessed during three assessments: at baseline, during second assessment ten weeks later, third assessment was carried out one year later
  To assess the impact of visual cues on handwriting, patients were instructed to write one simple and one complex sentence on white, striped and squared paper. During assessment, the speed of writing was registered.

OTHER OUTCOMES:
Quality of life: its change as a result of physiotherapy and change over time | it was assessed during all the assessments: at baseline, during second assessment ten weeks later, third assessment was carried out one year later, forth assessment was conducted another year later
  it was assessed with PDQ-39 questionaire
prevalence of pain: its change as a result of physiotherapy and change over time | it was assessed during all the assessments: at baseline, during second assessment ten weeks later, third assessment was carried out one year later, forth assessment was conducted another year later
  it was assessed with patient interview
patient-specific complaints:its change as a result of physiotherapy and change over time | it was assessed during all the assessments: at baseline, during second assessment ten weeks later, third assessment was carried out one year later, forth assessment was conducted another year later
  it was assessed with patient interview
difficulties in executing different activities of daily living: its change as a result of physiotherapy and change over time | it was assessed during all the assessments: at baseline, during second assessment ten weeks later, third assessment was carried out one year later, forth assessment was conducted another year later
  it was assessed with patient interview

CONTACTS AND LOCATIONS:
Overall Officials: Kadri Medijainen, MSc, Principal Investigator — Junior research fellow in physiotherapy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2024 Apr 8;4(4):CD013856. doi: 10.1002/14651858.CD013856.pub3. PMID 38588457
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Jan 5;1(1):CD013856. doi: 10.1002/14651858.CD013856.pub2. PMID 36602886